CLINICAL TRIAL: NCT01062425
Title: Randomized, Phase II, Double-Blind, Placebo-Controlled Trial of Conventional Chemoradiation and Adjuvant Temozolomide Plus Cediranib Versus Conventional Chemoradiation and Adjuvant Temozolomide Plus Placebo in Patients With Newly Diagnosed Glioblastoma
Brief Title: Temozolomide and Radiation Therapy With or Without Cediranib Maleate in Treating Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other); Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-02012; NCI-2011-02012 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000665163; RTOG-0837; RTOG 0837 (Other: NRG Oncology); RTOG-0837 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-05

CONDITIONS: Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy, Conformal; cediranib; Radiotherapy, Intensity-Modulated; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cediranib, TMZ, and RT (Experimental): Cediranib (3 days) followed by radiation therapy (RT) + daily temozolomide (TMZ) + cediranib followed by cediranib monotherapy (4 weeks) followed by TMZ + cediranib for 12 cycle maximum.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cediranib Maleate; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Temozolomide
- Placebo, TMZ, and RT (Active Comparator): Placebo (3 days) followed by radiation therapy (RT) + daily temozolomide (TMZ) + placebo followed by placebo monotherapy (4 weeks) followed by TMZ + placebo for 12 cycle maximum.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Drug: Temozolomide

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3-dimensional conformal radiotherapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
  Arms: Cediranib, TMZ, and RT
Radiation: Intensity-Modulated Radiation Therapy — Undergo intensity-modulated radiation therapy
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Placebo, TMZ, and RT
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This randomized phase II trial studies temozolomide, radiation therapy, and cediranib maleate to see how well they work compared with temozolomide, radiation therapy, and a placebo in treating patients with newly diagnosed glioblastoma (a type of brain tumor). Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x-rays to kill tumor cells. Cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether temozolomide and radiation therapy are more effective when given with or without cediranib maleate in treating glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the addition of cediranib (cediranib maleate) to chemoradiation treatment enhances treatment efficacy as measured by the 6-month progression-free survival rate.

SECONDARY OBJECTIVES:

I. To determine if the addition of cediranib to chemoradiation treatment enhances treatment efficacy as measured by overall survival.

II. To determine if the addition of cediranib to chemoradiation treatment enhances treatment efficacy as measured by progression-free survival.

III. To determine if there is an association between tumor O6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) gene methylation status and treatment response and outcome.

IV. To compare and record the toxicities of the cediranib + chemoradiation arm versus the chemoradiation arm.

V. To evaluate whether 6-month progression-free survival is associated with overall survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cediranib maleate orally (PO) once daily (QD) for 3 days. Patients then undergo radiation therapy (intensity-modulated radiation therapy or 3-dimensional conformal radiation therapy) QD, 5 days a week, for 6 weeks and receive temozolomide PO QD and cediranib maleate PO QD for 6 weeks. Patients then receive temozolomide PO QD alone on days 1-5. Treatment with temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO QD for 3 days. Patients then undergo radiation therapy (intensity-modulated radiation therapy or 3-dimensional conformal radiation therapy) QD, 5 days a week, for 6 weeks and receive temozolomide PO QD and placebo PO QD for 6 weeks. Patients then receive temozolomide PO QD alone on days 1-5. Treatment with temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of glioblastoma or gliosarcoma (World Health Organization [WHO] grade IV) confirmed by central review prior to step 2 registration
* Tumor tissue that is determined by central pathology review prior to step 2 registration to be of sufficient size for analysis of MGMT status

  * Patients must have at least 1 block of tumor tissue; submission of 2 blocks is strongly encouraged
  * Cavitron ultrasonic aspirator (CUSA)-derived material is not allowed; fresh frozen tumor tissue acquisition is encouraged
  * Diagnosis must be made by surgical excision, either partial or complete; stereotactic biopsy is not allowed because it will not provide sufficient tissue for MGMT analysis
  * The tumor tissue must be sent as soon as possible to maximize the likelihood of eligibility; tumor tissue may not be submitted later than 28 days after the surgical procedure, because tissue analysis will not be able to be performed in time for treatment to commence by the mandatory 6-week post-surgery outer limit; submission of tissue earlier than 28 days post-surgery is highly recommended
* The tumor must have a supratentorial component
* History/physical examination, including neurologic examination, within 14 days prior to step 2 registration
* The patient must have recovered from the effects of surgery, post-operative infection, and other complications before step 2 registration
* A diagnostic contrast-enhanced magnetic resonance imaging (MRI) of the brain must be performed preoperatively and postoperatively prior to step 1 registration; the postoperative scan must be performed within 28 days prior to step 1 registration
* Documentation of steroid doses/concurrent medications within 14 days prior to step 2 registration
* Karnofsky performance status >= 70 within 14 days prior to step 2 registration
* Complete blood count (CBC)/differential obtained within 14 days prior to step 2 registration on study, with adequate bone marrow function defined as follows:
* Absolute neutrophil count (ANC) >= 1,800 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >=10.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin (Hgb) >= 10.0 g/dl is acceptable)
* Adequate renal function, as defined below:
* Blood urea nitrogen (BUN) =< 30 mg/dl within 14 days prior to step 2 registration
* Creatinine =< 1.7 mg/dl within 14 days prior to step 2 registration
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 3 x normal range within 14 days prior to step 2 registration
* Systolic blood pressure =< 140 mm Hg AND diastolic pressure =< 90 mm Hg within 14 days prior to step 2 registration in the presence or absence of a stable regimen of anti-hypertensive therapy
* Prothrombin time/international normalized ratio (PT INR) < 1.4 for patients not on warfarin confirmed by testing within 1 week of step 2 registration
* Patients on full-dose anticoagulants (e.g., warfarin or low molecular weight [LMW] heparin) must meet both of the following criteria:

  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
  * In-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
* Patient must provide study specific informed consent prior to step 1 registration
* Women of childbearing potential and male participants must practice adequate contraception
* For females of child-bearing potential, negative serum pregnancy test within 14 days prior to step 2 registration

Exclusion Criteria:

* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for >= 3 years; (for example, carcinoma in situ of the breast, oral cavity, and cervix are all permissible)
* Recurrent or multifocal malignant gliomas
* Metastases detected below the tentorium or beyond the cranial vault
* Prior chemotherapy or radiosensitizers for cancers of the head and neck region; note that prior chemotherapy for a different cancer is allowable (except temozolomide or cediranib); prior use of Gliadel wafers or any other intratumoral or intracavitary treatment are not permitted
* Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization
  * Transmural myocardial infarction within the last 6 months
  * Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an electrocardiogram (EKG) performed within 14 days of step 2 registration
  * New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to step 2 registration
  * History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease
  * Evidence of bleeding diathesis or coagulopathy
  * Serious or non-healing wound, ulcer, or bone fracture or history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to step 2 registration, with the exception of the craniotomy for tumor resection
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of step 2 registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of step 2 registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol
  * Active connective tissue disorders, such as lupus or scleroderma, which in the opinion of the treating physician may put the patient at high risk for radiation toxicity
  * Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Pregnant or lactating women
* Prior allergic reaction to temozolomide
* Patients treated on any other therapeutic clinical protocols within 30 days prior to step 1 registration or during participation in the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib
* Mean QTc >500 msec (with Bazett's correction) in screening electrocardiogram or history of familial long QT syndrome or other significant ECG abnormality noted within 14 days of treatment
* Patients receiving concurrent vascular endothelial growth factor (VEGF) inhibitors are prohibited from participating in this study
* Patients must not be on enzyme-inducing anti-epileptic drugs (EIAED); patients may be on non-enzyme inducing anti-epileptic drugs (NEIAED) or may not be taking any anti-epileptic drugs; in patients who have previously been on EIAED there must be at least a 14 day period since the last dose of an EIAED before the first dose of cediranib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-02-26 (Actual); Primary Completion 2015-12-06 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy T Batchelor, Principal Investigator — NRG Oncology
Locations (105):
- United States (105):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - AdventHealth Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - University of Rochester, Rochester, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After patient registration, sites submitted tissue for central histology and methyltransferase (MGMT) gene methylation evaluation. If tissue was evaluable and a patient continued on study, then treatment arm was assigned. Two hundred sixty-one patients were registered, 103 did not continue to treatment assignment, 158 had treatment assigned.
Period: Overall Study
Arm/Group | Placebo, TMZ, and RT | Cediranib, TMZ, and RT
Started | 55 | 103
Completed | 52 (Randomized eligible subjects are considered to have completed the study.) | 97 (Randomized eligible subjects are considered to have completed the study.)
Not Completed | 3 | 6
Not completed — Protocol Violation | 3 | 6

BASELINE CHARACTERISTICS:
Population: All randomized and eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, TMZ, and RT | Cediranib, TMZ, and RT | Total
Number analyzed (Participants) | 52 | 97 | 149
Age, Continuous [Median (Full Range); unit: years] | 59 [37 to 82] | 61 [27 to 83] | 60 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 44 | 68
  Male | 28 | 53 | 81

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival Rate
Description: Six-month progression-free survival is the rate of patients who have NOT progressed at six months, where progressive disease is defined as any of the following: ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions; any new lesion; or clinical deterioration. Progression will be determined by central review of MRI exams, assessed using MacDonald criteria for progression versus response on 2D T1 and T2 weighted images.
Time Frame: From randomization to 6 months.
Population: Randomized eligible patients with evaluable data at six months. (From the randomized eligible patients, 2 patients withdrew prior to 6 months and 1 did not have an evaluable scan on the placebo arm, while 4 withdrew before 6 months, 3 did not have an evaluable scan, and 2 did not receive protocol treatment on the cediranib arm.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo, TMZ, and RT | Cediranib, TMZ, and RT
Number analyzed (Participants) | 49 | 88
percentage of participants | 24.5 [12.5 to 36.5] | 46.6 [36.2 to 57]
Statistical Analysis 1: Comparison: Placebo, TMZ, and RT vs Cediranib, TMZ, and RT; The null hypothesis was that the 6m PFS rates for both arms are 50%, and the alternative hypothesis was that patients receiving the experimental regimen would have a 6-month PFS rate of 66%. With 150 eligible patients, there would be an 80% statistical power to detect the 16% absolute increase in 6m PFS at a significance level of 0.15, using a one-sided Z test for two proportions; Test type: Superiority or Other; p = 0.005, Z-test — One-sided test with significance level of 0.15

2. Secondary Outcome: Overall Survival (OS)
Description: OS will be estimated using the Kaplan-Meier method and differences between treatment arms will be tested using the log rank test. Multivariate analyses with the Cox proportional hazard model for OS will be performed with the stratification variables as fixed variables to assess the treatment effect adjusting patient-specific risk factors.
Time Frame: From randomization to time of death due to any cause. Patients are followed until death. Analysis occurs after all patients have been potentially followed for six months.
Population: All randomized and eligible patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo, TMZ, and RT | Cediranib, TMZ, and RT
Number analyzed (Participants) | 52 | 97
Months | 13.8 [9.6 to 18.9] | 14.5 [12.3 to 19.7]
Statistical Analysis 1: Comparison: Placebo, TMZ, and RT vs Cediranib, TMZ, and RT; Test type: Superiority or Other; p = 0.44, Log Rank — Significance level 0.05, two-sided test; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.6 to 1.24] — Placebo is the reference arm for the hazard ratio
Statistical Analysis 2: Comparison: Placebo, TMZ, and RT vs Cediranib, TMZ, and RT; Multivariate analysis with the Cox proportional hazard model for overall survival was performed with the stratification variables as fixed variables to assess the treatment effect adjusting patient-specific risk factors. The covariates evaluated for the multivariate models were assigned protocol treatment, MGMT methylation status, and RPA risk class; Test type: Superiority or Other; p = 0.648, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.62 to 1.34] — Placebo is reference level for the hazard ratio

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival time is defined as time from randomization to date of first progression or death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive without progression are censored at the date of last contact. Progression is defined as any of the following: ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions; any new lesion; or clinical deterioration.
Time Frame: From randomization to time of first progression or death due to any cause. Patients are followed until death. Analysis occurs after all patients have been potentially followed for six months.
Population: All randomized and eligible patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo, TMZ, and RT | Cediranib, TMZ, and RT
Number analyzed (Participants) | 52 | 97
Months | 2.7 [2.5 to 3.7] | 6.2 [4.5 to 8.1]
Statistical Analysis 1: Comparison: Placebo, TMZ, and RT vs Cediranib, TMZ, and RT; Test type: Superiority or Other; p = 0.03, Log Rank — Significance level 0.05, two-sided test; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.47 to 0.95] — Placebo is the reference arm for the hazard ratio
Statistical Analysis 2: Comparison: Placebo, TMZ, and RT vs Cediranib, TMZ, and RT; Multivariate analysis with the Cox proportional hazard model for progression-free survival was performed with the stratification variables as fixed variables to assess the treatment effect adjusting patient-specific risk factors. The covariates evaluated for the multivariate models were assigned protocol treatment, MGMT methylation status, and recursive partitioning analysis (RPA) risk class; Test type: Superiority or Other; p = 0.036, Regression, Cox; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.46 to 0.97] — Placebo is the reference arm

4. Secondary Outcome: Incidence of Grade 3+ Toxicities
Description: The number of patients with reported grade 3 and higher treatment-related toxicities as assessed by Common Terminology Criteria for Adverse Events version 4.0
Time Frame: From randomization to six months.
Population: All randomized and eligible patients who started protocol treatment.
Measure: Number; unit: participants
Arm/Group | Placebo, TMZ, and RT | Cediranib, TMZ, and RT
Number analyzed (Participants) | 52 | 92
participants | 35 | 77
Statistical Analysis 1: Comparison: Placebo, TMZ, and RT vs Cediranib, TMZ, and RT; Test type: Superiority or Other; p = 0.02, Chi-squared — Significance level 0.05, two-sided test

ADVERSE EVENTS:
Time Frame: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events (AE).
Description: All randomized and eligible patients who started protocol treatment.
Arm/Group | Placebo, TMZ, and RT | Cediranib, TMZ, and RT
Serious Adverse Events (participants affected / at risk) | 23/52 | 53/92
Other Adverse Events (participants affected / at risk) | 49/52 | 88/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo, TMZ, and RT (N=52) | Cediranib, TMZ, and RT (N=92)
Anemia (Blood and lymphatic system disorders) | 3 | 4
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 1
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 4
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Chills (General disorders) | 0 | 1
Death NOS (General disorders) | 2 | 1
Edema limbs (General disorders) | 1 | 2
Fatigue (General disorders) | 3 | 6
Fever (General disorders) | 0 | 2
Gait disturbance (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Bladder infection (Infections and infestations) | 0 | 1
Encephalomyelitis infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 2 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Soft tissue infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Wound infection (Infections and infestations) | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 5
Neutrophil count decreased (Investigations) | 2 | 8
Platelet count decreased (Investigations) | 3 | 17
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 9
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 6
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Ataxia (Nervous system disorders) | 1 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 2
Concentration impairment (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Hydrocephalus (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 1 | 3
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 5 | 8
Somnolence (Nervous system disorders) | 1 | 1
Stroke (Nervous system disorders) | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 2
Hallucinations (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 2
Thromboembolic event (Vascular disorders) | 5 | 5
Vascular disorders - Other (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo, TMZ, and RT (N=52) | Cediranib, TMZ, and RT (N=92)
Anemia (Blood and lymphatic system disorders) | 20 | 27
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 5 | 4
Ear pain (Ear and labyrinth disorders) | 3 | 2
Hearing impaired (Ear and labyrinth disorders) | 3 | 2
Tinnitus (Ear and labyrinth disorders) | 3 | 6
Hypothyroidism (Endocrine disorders) | 0 | 6
Blurred vision (Eye disorders) | 3 | 13
Eye disorders - Other (Eye disorders) | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 18
Constipation (Gastrointestinal disorders) | 24 | 41
Diarrhea (Gastrointestinal disorders) | 8 | 53
Dry mouth (Gastrointestinal disorders) | 1 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 7
Dysphagia (Gastrointestinal disorders) | 1 | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 6
Mucositis oral (Gastrointestinal disorders) | 0 | 6
Nausea (Gastrointestinal disorders) | 20 | 59
Vomiting (Gastrointestinal disorders) | 4 | 30
Chills (General disorders) | 1 | 6
Edema face (General disorders) | 6 | 3
Edema limbs (General disorders) | 5 | 7
Fatigue (General disorders) | 41 | 77
Fever (General disorders) | 3 | 7
Gait disturbance (General disorders) | 8 | 8
Malaise (General disorders) | 0 | 5
Pain (General disorders) | 3 | 6
Mucosal infection (Infections and infestations) | 4 | 9
Urinary tract infection (Infections and infestations) | 5 | 6
Bruising (Injury, poisoning and procedural complications) | 0 | 7
Dermatitis radiation (Injury, poisoning and procedural complications) | 10 | 15
Fall (Injury, poisoning and procedural complications) | 3 | 5
Alanine aminotransferase increased (Investigations) | 14 | 41
Alkaline phosphatase increased (Investigations) | 2 | 8
Aspartate aminotransferase increased (Investigations) | 6 | 25
Blood bilirubin increased (Investigations) | 3 | 10
CD4 lymphocytes decreased (Investigations) | 3 | 3
Creatinine increased (Investigations) | 5 | 16
Hemoglobin increased (Investigations) | 1 | 6
Investigations - Other (Investigations) | 10 | 21
Lymphocyte count decreased (Investigations) | 17 | 35
Neutrophil count decreased (Investigations) | 7 | 25
Platelet count decreased (Investigations) | 19 | 54
Weight loss (Investigations) | 6 | 24
White blood cell decreased (Investigations) | 14 | 40
Anorexia (Metabolism and nutrition disorders) | 22 | 42
Dehydration (Metabolism and nutrition disorders) | 2 | 13
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 19 | 35
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 11
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 8
Hypernatremia (Metabolism and nutrition disorders) | 6 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 15
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 21
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 6
Hypokalemia (Metabolism and nutrition disorders) | 12 | 18
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 8
Hyponatremia (Metabolism and nutrition disorders) | 11 | 27
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 8
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 7 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 | 23
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3 | 3
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 10
Amnesia (Nervous system disorders) | 4 | 2
Ataxia (Nervous system disorders) | 7 | 15
Cognitive disturbance (Nervous system disorders) | 4 | 7
Dizziness (Nervous system disorders) | 14 | 25
Dysarthria (Nervous system disorders) | 1 | 5
Dysgeusia (Nervous system disorders) | 12 | 20
Dysphasia (Nervous system disorders) | 4 | 14
Facial muscle weakness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 27 | 48
Memory impairment (Nervous system disorders) | 13 | 13
Nervous system disorders - Other (Nervous system disorders) | 2 | 11
Paresthesia (Nervous system disorders) | 3 | 4
Peripheral motor neuropathy (Nervous system disorders) | 5 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 9
Seizure (Nervous system disorders) | 4 | 15
Somnolence (Nervous system disorders) | 3 | 4
Tremor (Nervous system disorders) | 4 | 4
Agitation (Psychiatric disorders) | 3 | 5
Anxiety (Psychiatric disorders) | 8 | 15
Confusion (Psychiatric disorders) | 6 | 9
Depression (Psychiatric disorders) | 3 | 14
Insomnia (Psychiatric disorders) | 11 | 20
Personality change (Psychiatric disorders) | 3 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 47
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 12
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 10
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 6
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 6 | 12
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 5
Hypertension (Vascular disorders) | 8 | 32
Hypotension (Vascular disorders) | 3 | 5
Thromboembolic event (Vascular disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.